CLINICAL TRIAL: NCT06591650
Title: A Phase II Study of Gemcitabine, Cisplatin, Nab-Paclitaxel, and Durvalumab in Locally Advanced or Metastatic Gallbladder Cancer
Brief Title: Gemcitabine Hydrochloride, Cisplatin, Nab-Paclitaxel, and Durvalumab in Treating Patients with Locally Advanced or Metastatic Gallbladder Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lunxiu Qin, vice president of hospital, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Huashan010
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Gallbladder Cancer Unresectable
MeSH Terms: interventions — Gemcitabine; Cisplatin; 130-nm albumin-bound paclitaxel; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Gemcitabine + Cisplatin + Nab-Paclitaxel + Durvalumab (Experimental): Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes, cisplatin IV over 60 minutes and nab-paclitaxel over 30 minutes on days 1 and 8. Durvalumab intravenously (IV) on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gemcitabine hydrochloride; Drug: Cisplatin; Drug: Nab-paclitaxel; Drug: Durvalumab

INTERVENTIONS:
Drug: gemcitabine hydrochloride — 800 mg/m^2, intravenous (IV) over 30 minutes, Days 1,8, every 21 days.
Drug: Cisplatin — 25 mg/m^2, intravenous (IV) over 60 minutes, Days 1,8, every 21 days.
Drug: Nab-paclitaxel — 100 mg/m^2, intravenous (IV) over 30 minutes, Days 1,8, every 21 days.
Drug: Durvalumab — 1500mg, intravenous (IV) over 30 minutes, Days 1, every 21 days.

SUMMARY:
This phase II trail will evaluate the efficacy and safety of combining gemcitabine hydrochloride, cisplatin, nab-paclitaxel (paclitaxel albumin-stabilized nanoparticle formulation), with durvalumab in treating patients who have locally advanced or metastatic gallbladder cancer.

Drugs used in chemotherapy, such as gemcitabine hydrochloride, cisplatin, and nab-paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Durvalumab is a type of drug called a monoclonal antibody, which selectively blocks PD-L1 binding to PD-1. This anti-PD-L1 treatment works by allowing the immune system to detect your cancer and reactivates the immune response.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years at time of study entry.
2. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
3. Has histologically or cytologically confirmed unresectable locally advanced or metastatic gallbladder adenocarcinoma.
4. Has at least 1 measurable disease, as defined by RECIST 1.1, at baseline.
5. Has a life expectancy ≥ 3 months from proposed first dose date.
6. Has received no prior anti-cancer therapy for gallbladder adenocarcinoma.
7. Has adequate bone marrow, liver and renal functions measured within 14 days prior to administration of study treatment: Absolute neutrophil count≥1.5 x109/L;Platelet count≥100×109/L;Serum bilirubin≤2.5×institutional upper limit of normal (ULN). Subjects requiring biliary decompression, biliary stent, or drainage using percutaneous trans-hepatic cholangiogram are allowed (patients with a declining bilirubin status post stent placement are eligible with serum bilirubin≤2.5×ULN);Aspartate aminotransferase (AST)/alanine aminotransferase (ALT)≤2.5×ULN;Measured creatinine clearance (CL)>50 mL/min or calculated creatinine CL> 50 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.
8. Women with childbearing potential should complete a pregnancy test with negative result within 28 days of study treatment and be willing to use effective contraceptive methods from screening to 90 days after the last dose of durvalumab
9. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm from screening to 90 days after the last dose of durvalumab.
10. Capable of giving written informed consent, prior to any study specific procedures,and ability to comply with the study protocol in the investigator's judgment.

Exclusion Criteria:

1. Diagnosis of intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma or carcinoma of Vaters ampulla.
2. Known hypersensitivity to any of the study drugs or any of the study drug excipients.
3. Patients, who have received prior anti-PD-1, anti PD-L1 or anti CTLA-4 therapy.
4. Has an active or previously documented autoimmune or inflammatory disorder (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [diverticulosis is not an excluding factor], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]).
5. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable: Patients with vitiligo or alopecia; Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement; Patients having any chronic skin condition that does not require systemic therapy; Patients without active disease in the last 5 years (allowed only after consultation with the study physician); Patients with celiac disease controlled by diet alone.
6. Has history of allogenic organ transplantation.
7. Has a history of active primary immunodeficiency.
8. Has uncontrolled intercurrent illness, including but not limited to, ongoing or active infection; symptomatic congestive heart failure; uncontrolled hypertension; unstable angina pectoris; cardiac arrhythmia; interstitial lung disease; serious chronic gastrointestinal conditions associated with diarrhea; or psychiatric illness/social situations that would limit compliance with study requirements, would substantially increase risk of incurring adverse events (AEs), or would compromise the ability of the patient to give written informed consent.
9. Has a prior history of myocardial infarction, transient ischemic attack, or stroke within the past 3 months prior to the scheduled first dose of study treatment.
10. Has a history of another primary malignancy. Patients having the following are still eligible: Malignancy treated with curative intent, no known active disease >= 5 years before the first dose of IP, and low potential risk for recurrence; Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; Adequately treated carcinoma in situ without evidence of disease.
11. Has active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis [TB] testing in line with local practice), hepatitis B (presence of hepatitis B surface antigen [HBsAg] and/or anti-HBcAb with detectable hepatitis B virus [HBV] DNA ≥10 IU/mL), or hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (hepatitis C virus [HCV]) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA).
12. Is currently using or previously used immunosuppressive medication within 14 days before the first dose of durvalumab. The following medications are exceptions to this criterion: Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection); Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent; Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication).
13. Is a female and pregnant or breastfeeding; or is a male or female of reproductive potential who is not willing to employ effective birth control from time of screening to 90 days after the last dose of durvalumab.
14. Participated in another clinical study with an investigational product during the last 4 weeks from the first dose of this study's treatment.
15. Is concurrently enrolled in another clinical study (patient is eligible if the study is an observational (non interventional) study or if enrollment is during the follow-up period of an interventional study.
16. Is unsuitable to participate in the study or is unlikely to comply with study procedures, restrictions and requirements (per judgment by the investigator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Tumor assessments (per RECIST 1.1) every 6 weeks for the first 24 weeks relative to the date of randomization and then every 8 weeks thereafter. Assessed up to maximum of approximately 36 months.
  Disease assessments based on investigator assessments were determined by using RECIST version 1.1 guidelines. The ORR was defined as the percentage of patients with confirmed complete response (CR) or confirmed partial response (PR). The CR was defined as disappearance of all target and non-target lesions and no new lesions. The PR was defined as ≥ 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new non-target lesion. A confirmed CR or PR was defined as 2 CRs or 2 PRs with no evidence of progression in-between. Patients who discontinued randomized treatment without progression, received a subsequent anti-cancer therapy and then responded were not included as responders for ORR.

SECONDARY OUTCOMES:
Progressive-free survival (PFS) | Tumor assessments every 6 weeks after treatment for the first 24 weeks and then every 8 weeks thereafter until date of RECIST 1.1 defined radiological progressive disease or death. Assessed up to maximum of approximately 36 months.
  PFS based on investigator assessments according to RECIST version 1.1 was defined as time from date of treatment until date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdrew from therapy or received another anticancer therapy prior to progression. Progression (i.e., PD) was defined as at least a 20% increase in the sum of diameters of target lesions (TLs) and an absolute increase of ≥ 5mm, taking as reference the smallest sum of diameters since treatment started including the baseline sum of diameters, or a measurable increase in a non-target lesion, or the appearance of new lesions. Median PFS was calculated using the Kaplan-Meier technique.
Overall Survival (OS) | From date of treatment until death due to any cause. Assessed up to maximum of approximately 36 months.
  Overall Survival (OS) was defined as the time from the date of treatment until death due to any cause. Any patient not known to have died at the time of analysis was censored based on the last recorded date on which the patient was known to be alive. Median OS was calculated using the Kaplan-Meier technique.
Duration of Response (DoR) | Tumor assessments (per RECIST 1.1) every 6 weeks for first 24 weeks relative to the date of treatment and then every 8 weeks thereafter. Assessed up to maximum of approximately 36 months.
  The DoR was defined as the time from the date of first documented OR (confirmed CR or confirmed PR) until date of documented progression (PD) based on investigator assessments by using RECIST version 1.1 or death in absence of disease progression. A confirmed CR was defined in above outcome measures. The PD was defined at least 20% increase in sum of diameters of target lesions, unequivocal progression of existing non-target lesions or new lesion. For participants who were alive and no documented PD at the time of data cutoff for analysis, DoR was censored at the last evaluable disease assessment date. Median DoR was calculated using Kaplan-Meier method.
Disease Control Rate (DCR) | Tumor assessments (per RECIST 1.1) every 6 weeks for the first 24 weeks relative to the date of treatment and then every 8 weeks thereafter. Assessed up to maximum of approximately 36 months.
  Disease control rate based on investigator assessments according to RECIST version 1.1 was defined as the rate of best objective response of complete response (CR), partial response (PR) or stable disease (SD).

CONTACTS AND LOCATIONS:
Overall Officials: Lun xiu Qin, Principal Investigator — Fudan University
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China